CLINICAL TRIAL: NCT04048330
Title: Periconceptional Surveillance for Prevention of Anemia and Birth Defects in India
Brief Title: Periconceptional Surveillance in India
Status: Active, not recruiting | Type: Observational
Sponsor: Cornell University (Other)
Collaborators: Arogyavaram Medical Centre (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); St. John's Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 76461
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Anemia; Folate Deficiency; Vitamin B12 Deficiency
Keywords: Anemia; Periconceptional; Vitamin B12; Folate; Surveillance; India
MeSH Terms: conditions — Anemia; Folic Acid Deficiency; Vitamin B 12 Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological specimens collected will include archived blood, saliva, urine, and stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women of reproductive age: Women 15 to 49 years of age who are not pregnant or lactating

SUMMARY:
Women of reproductive age are a high-risk population for anaemia and micronutrient deficiencies. Evidence supports the role of periconceptional nutrition in the development of adverse pregnancy complications. However, in India, there are limited population-based data to guide evidence-based recommendations and priority setting. The objective of this study is to conduct a population-based biomarker survey of anaemia and vitamin B12 and folate status in women of reproductive age as part of a periconceptional surveillance program in Southern India.

DETAILED DESCRIPTION:
Women of reproductive age are a high-risk population for anemia and micronutrient deficiencies due to social structures, and the physical demands of pregnancy and lactation particularly in South Asia. Inadequate periconceptional folate and vitamin B12 status are implicated in the development of birth defects and other pregnancy complications. Randomized trials established that periconceptional folic acid supplementation can prevent the occurrence and recurrence of neural tube defects, and fortification of staple foods with folic acid has been associated with decreasing neural tube defects in many countries around the globe. Red blood cell folate has been identified as a biomarker of neural tube defect risk at the population level, and increases in RBC folate concentrations predicted reductions in neural tube defect risk of up to 10-fold in USA, Chinese and Irish populations.

Emerging evidence has identified maternal vitamin B12 deficiency as a risk factor for neural tube defects, and vitamin B12 status may modify circulating folate biomarkers that predict neural tube defect risk. It is estimated that the burden of neural tube defects in India is among the highest in the world. However, there is little representative population-level data from Southern India. Surveillance programs are urgently needed to establish the burden of anaemia and key micronutrient deficiencies in settings such as Southern India to inform interventions for anemia and birth defects prevention.

The objective of this study is to conduct a biomarker survey of anemia and vitamin B12 and folate status in women of reproductive age as part of a periconceptional surveillance program in Southern India and to inform the development of a randomized trial for anemia and birth defects prevention. As part of this surveillance program, we are also establishing the World Health Organization-recommended microbiological assay for folate at our laboratory in Bangalore, India, and a WHO-SEARO site for birth defects surveillance in this setting. Findings from this pre-intervention biomarker survey will directly inform the development of a randomized efficacy trial of quadruple-fortified salt for the prevention of anemia and birth defects in Southern India and serve as the foundation for future public health programs to improve the health of women and young children in this population.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 15 to 49 years
* Currently not pregnant or lactating

Exclusion Criteria:

* <15 or >49 years old
* Currently pregnant or lactating

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: In order to obtain representative, population-level data in this setting, all rural households and a random subset of urban households in the catchment area will be selected for subsequent screening and recruitment of women for the biomarker study, with a target sample size of 2,000 women of reproductive age.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-04-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | Baseline
  Hemoglobin concentrations, g/dL
Folate status | Baseline
  Erythrocyte and serum folate concentrations, nmol/L
Vitamin B12 status | Baseline
  Total vitamin B12 concentrations, pmol/L

SECONDARY OUTCOMES:
Anemia | Baseline
  Hemoglobin <12.0 g/dL
Folate deficiency and insufficiency | Baseline
  Erythrocyte (RBC) folate <305 nmol/L; <748 nmol/L
Vitamin B12 deficiency and insufficiency | Baseline
  Total vitamin B12 <148 pmol/L; <221 pmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Julia L Finkelstein, MPH SM ScD, Principal Investigator — Cornell University
Locations (1):
- Arogyavaram Medical Centre, Madanapalle, Andhra Pradesh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finkelstein JL, Fothergill A, Johnson CB, Guetterman HM, Bose B, Jabbar S, Zhang M, Pfeiffer CM, Qi YP, Rose CE, Krisher JT, Ruth CJ, Mehta R, Williams JL, Bonam W, Crider KS. Periconceptional surveillance for prevention of anaemia and birth defects in Southern India: protocol for a biomarker survey in women of reproductive age. BMJ Open. 2020 Oct 29;10(10):e038305. doi: 10.1136/bmjopen-2020-038305. PMID 33122315
- [Result] Finkelstein JL, Fothergill A, Johnson CB, Guetterman HM, Bose B, Jabbar S, Zhang M, Pfeiffer CM, Qi YP, Rose CE, Williams JL, Bonam W, Crider KS. Anemia and Vitamin B-12 and Folate Status in Women of Reproductive Age in Southern India: Estimating Population-Based Risk of Neural Tube Defects. Curr Dev Nutr. 2021 Apr 26;5(5):nzab069. doi: 10.1093/cdn/nzab069. eCollection 2021 May. PMID 34027296
- [Result] Finkelstein JL, Fothergill A, Guetterman HM, Johnson CB, Bose B, Qi YP, Rose CE, Williams JL, Mehta S, Kuriyan R, Bonam W, Crider KS. Iron status and inflammation in women of reproductive age: A population-based biomarker survey and clinical study. Clin Nutr ESPEN. 2022 Jun;49:483-494. doi: 10.1016/j.clnesp.2022.02.123. Epub 2022 Mar 5. PMID 35623855
- [Result] Fothergill A, Crider KS, Johnson CB, Raj MP, Guetterman HM, Bose B, Rose CE, Qi YP, Williams JL, Kuriyan R, Bonam W, Finkelstein JL. Comparison of Anemia Screening Methods Using Paired Venous Samples in Women of Reproductive Age in Southern India. J Nutr. 2023 Jan 14;152(12):2978-2992. doi: 10.1093/jn/nxac218. PMID 36130238
- [Result] Fothergill A, Crider KS, Rose CE, Bose B, Guetterman HM, Johnson CB, Jabbar S, Zhang M, Pfeiffer CM, Qi YP, Williams JL, Kuriyan R, Bonam W, Finkelstein JL. Estimating the serum folate concentration that corresponds to the red blood cell folate concentration threshold associated with optimal neural tube defects prevention: A population-based biomarker survey in Southern India. Am J Clin Nutr. 2023 May;117(5):985-997. doi: 10.1016/j.ajcnut.2023.01.016. Epub 2023 Apr 19. PMID 37137617
- [Derived] Guetterman HM, Crider KS, Fothergill A, Bose B, Johnson CB, Jabbar S, Zhang M, Pfeiffer CM, Rose CE, Qi YP, Williams JL, Mehta S, Kuriyan R, Finkelstein JL. Vitamin B12 status and metabolic health in women of reproductive age: Population-based biomarker survey. Clin Nutr ESPEN. 2025 Aug;68:176-188. doi: 10.1016/j.clnesp.2025.05.011. Epub 2025 May 9. PMID 40349845